CLINICAL TRIAL: NCT01263171
Title: A Stratified Phase II Study of Neoadjuvant Chemotherapy Given Before SCPRT as Treatment for Patients With MRI-Staged Operable Rectal Cancer at High Risk of Metastatic Relapse
Brief Title: Oxaliplatin, Leucovorin, and Fluorouracil Before and After Radiation Therapy and Surgery in Treating Patients With Rectal Cancer That Can Be Removed by Surgery
Acronym: COPERNICUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cardiff University (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000691166; WCTU-COPERNICUS (Other: Cardiff University); 2010-023083-40 (EudraCT Number); C23134/A11537 (Other Grant/Funding Number: Cancer Research UK); CARDIFF-SPON830-10 (Other: Cardiff University)
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage IIIB rectal cancer; stage IIIC rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Leucovorin; Fluorouracil; Oxaliplatin; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neo-adjuvant chemotherapy (Other): Neo-adjuvant chemotherapy prior to short course pre-operative radiotherapy followed by adjuvant chemotherapy.
  Interventions: Drug: Leucovorin; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: Leucovorin
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, leucovorin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying giving oxaliplatin, leucovorin, and fluorouracil together, before and after radiation therapy and surgery in treating patients with rectal cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the feasibility of introducing 8 weeks of neoadjuvant oxaliplatin and fluorouracil followed by radiotherapy and immediate surgical resection in patients with resectable adenocarcinoma of the rectum.

Secondary

* Determine feasibility of achieving dose intensity for chemotherapy and radiotherapy in these patients.
* Determine the safety, in terms of NCI CTCAE version 4 toxicities, including postoperative complication rate (up to 30 days postoperatively), and late toxicity assessment at 1 year following surgery, in these patients.
* Determine how active is the neoadjuvant chemotherapy, in terms of down staging the rectal cancer, local recurrence-free, distant metastasis-free, and overall survival at 1 year following surgery in these patients.

Neoadjuvant therapy: Patients receive oxaliplatin and leucovorin (L-leucovorin or leucovorin calcium) IV over 2 hours on day 1 and fluorouracil IV over 46 hours on days 1-2. Treatment repeats every 2 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Radiotherapy/Surgery: Beginning 1 week after completion of chemotherapy, patients undergo radiotherapy, followed by surgical resection of their primary tumor, within 7-14 days after completion of radiotherapy. Between 6-8 weeks following surgery, patients begin adjuvant therapy.

Adjuvant therapy: Patients receive oxaliplatin and leucovorin (L-leucovorin or leucovorin calcium) IV over 2 hours on day 1 and fluorouracil IV over 46 hours on days 1-2. Treatment repeats every 2 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Blood and biopsy specimens are collected at baseline and periodically for translational research studies.

After completion of study therapy, patients are followed up periodically for 1 year.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histopathologically confirmed rectal adenocarcinoma meeting the following criteria:

  * Inferior aspect of tumor is > 4 cm from anal verge on digital examination and pelvic MRI scan
  * Superior aspect of tumor is not higher than the anterior aspect of the S1/S2 interspace on pelvic MRI scan
  * Mesorectal fascia is not threatened or involved (tumor > 1 mm from mesorectal fascia)
  * Primary tumor meets 1 of the following criteria:

    * T3a-b (mesorectal primary tumor invasion seen ≤ 5 mm beyond muscularis propria) in the presence of 1 of the following:

      * Extra-mural vascular invasion
      * Mesorectal lymph node(s)/tumor deposit(s) with irregular border and mixed signal intensity
    * Any T3c (primary tumor invasion seen > 5 mm beyond muscularis propria)-T4a (invasion of visceral peritoneum for tumors with a component above peritoneal reflection)
  * Low tumors should not involve levator ani (> 1 mm gap between tumor and levator ani) or anal sphincters
* No evidence of distant metastases or stage T4b cancer with invasion into adjacent organs or structures
* Must have measurable disease at the baseline visit
* Impending rectal obstruction is permitted if relieved by a non-functioning ileostomy or colostomy
* No disease threatening mesorectal fascia (disease ≤ 1 mm from mesorectal fascia whether this is primary tumor, extra-mural vascular invasion, or tumor deposit with irregular border and mixed signal intensity)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Hemoglobin ≥ 9 g/dL
* WBC ≥ 3 x 10^9/L
* Absolute neutrophil count ≥ 1.5 x10^9/L
* Platelet count ≥ 100 x10^9/L
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 x ULN
* AST or ALT ≤ 2.5 x ULN
* Creatinine clearance ≥ 50 mL/min
* Magnesium and calcium normal
* Candidate for systemic therapy, in the opinion of the primary oncologist
* No known significant impairment of intestinal absorption (e.g., chronic diarrhea, inflammatory bowel disease)
* No evidence of established or acute ischemic heart disease (e.g., left bundle branch block, pathological q-waves, ST elevation, or ST-segment depression) and normal clinical cardiovascular assessment by ECG
* No enlarged pelvic sidewall lymph nodes
* No severe local bowel symptoms of tenesmus or irregularity or frequency of bowel habit precluding accurate assessment of diarrhea
* No pelvic sepsis
* No uncontrolled infection
* Not pregnant or nursing
* Fertile patients must use effective contraception during treatment and for 6 months after completion of treatment
* No other prior or current malignant disease that, in the judgement of the treating investigator, is likely to interfere with study treatment or assessment of response
* No clinically significant cardiovascular disease, including any of the following within the past year:

  * Myocardial infarction
  * Unstable angina
  * Symptomatic congestive heart failure
  * Serious uncontrolled cardiac arrhythmia
* No history of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease)

PRIOR CONCURRENT THERAPY:

* No prior pelvic radiotherapy
* No metallic colon stent or rectal stent in situ
* More than 30 days since prior chemotherapy, radiotherapy, hormonal treatment, antibody therapy, immunotherapy, gene therapy, vaccine therapy, angiogenesis inhibitors, matrix metalloproteinase inhibitors, thalidomide, anti-VEGF/Flk-1 monoclonal antibodies, or other experimental drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who commence neoadjuvant chemotherapy and radiotherapy and then undergo surgical resection | Two years

SECONDARY OUTCOMES:
Feasibility in terms of achieved dose intensity for chemotherapy and radiotherapy | Two years
Safety in terms of NCI CTCAE v 4 toxicities up to 30 days postoperatively and late toxicity at 1 year after surgery | Two years
Complete response | Two years
Efficacy in terms of down-staging rectal cancer | Two years
Local recurrence-free, distant metastasis-free, and overall survival at 1 year after surgery | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Simon Gollins, MD, Principal Investigator — Glan Clwyd Hospital
Locations (7):
- United Kingdom (7):
  - Walsgrave Hospital, Coventry, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Christie Hospital, Manchester, England
  - Rosemere Cancer Centre at Royal Preston Hospital, Preston, England
  - Royal Marsden - Surrey, Sutton, England
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales

IPD SHARING:
Plan to Share IPD: Undecided